CLINICAL TRIAL: NCT05571345
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled Crossover Study to Evaluate the Oral Abuse Potential of PF614 Compared with Oxycodone Immediate-Release Tablets and Placebo in Non-Dependent Recreational Opioid Users
Brief Title: A Study to Evaluate the Oral Abuse Potential of PF614 in Non-Dependent Recreational Opioid Users (PF614-104)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ensysce Biosciences (Industry)
Collaborators: Dr. Vince Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PF614-104
Record Dates: First submitted 2022-09-15; First posted 2022-10-07 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Recreational Drug Use
Keywords: Non-dependent
MeSH Terms: conditions — Recreational Drug Use | interventions — Oxycodone; Tablets

STUDY DESIGN:
Intervention Model Description: The Treatment Phase will consist of 5 treatment periods. Subjects will receive each of the following 5 treatments (1 per treatment period) in a randomized, double-blind, crossover manner, following a fasting period of at least 8 hours. Pharmacodynamic, pharmacokinetic and safety assessments will be conducted prior to dosing and for 24 hours after each study drug administration. Each study drug administration will be separated by a washout interval of approximately 120 hours. All subjects will remain in clinic for the duration of the Treatment Phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will involve 2 double-blind phases. Within each of the double-blind Qualification and Treatment Phases, treatments will be matched in appearance and subjects will ingest the same number of oral capsules in each treatment period.
  Neither the subject nor the blinded site personnel will know which treatment is being administered to each subject during the double-blind Qualification and Treatment Phases.
  In the Treatment Phase, under normal circumstances, the blind will not be broken until all subjects have completed treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- PF614 50 mg (Experimental): PF614 50 mg capsule (1 x 50 mg capsule over-encapsulated and 1 x placebo to match PF614 capsule)
  Interventions: Drug: PF614
- PF614 100 mg (Experimental): PF614 100 mg capsule (1 x 100 mg capsule and 1 x placebo to match PF614 capsule)
  Interventions: Drug: PF614
- PF614 200 mg (Experimental): PF614 200 mg capsule (2 x 100 mg capsules)
  Interventions: Drug: PF614
- Oxycodone IR 40 mg (Active Comparator): Oxycodone HCl 40 mg (2 x 20 mg capsules over-encapsulated to match PF614 capsules).
  Interventions: Drug: Oxycodone Hydrochloride 40 mg
- Placebo (Placebo Comparator): Placebo capsules to match PF614 (2 x placebo capsules)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF614 — PF614 capsules (50 mg or 100 mg)
  Other Names: Oxycodone prodrug
  Arms: PF614 100 mg; PF614 200 mg; PF614 50 mg
Drug: Oxycodone Hydrochloride 40 mg — Oral 20 mg tablets (two each)
  Other Names: Oxycodone hydrochloride (HCl) immediate-release (IR) tablets, 40 mg; Roxicodone or generic equivalent, 40 mg
  Arms: Oxycodone IR 40 mg
Drug: Placebo — Placebo to match PF614 capsules will be provided by the sponsor.
  Other Names: Placebo capsules
  Arms: Placebo

SUMMARY:
This will be a randomized, double-blind, placebo- and active-controlled, 5-way crossover study to evaluate the abuse potential, safety and pharmacokinetics of orally administered PF614 relative to oxycodone IR (immediate-release) tablets and placebo.

DETAILED DESCRIPTION:
The study will consist of 4 phases: Screening, Qualification, Treatment and Follow-up.

1. Screening Visit (Visit 1) The Screening Phase will be completed as an outpatient visit within 28 days of the Qualification Phase and will consist of a standard medical screen.
2. Qualification Phase (Visit 2) Within 28 days of a standard medical screening, eligible subjects will return to the clinical site as inpatients to complete the Qualification Phase (Visit 2). Upon admission to the clinical site, subjects will be interviewed and assessed for continued eligibility for the study. Subjects will check into the inpatient facility on Day -1.

   The Qualification Phase will include a Naloxone Challenge Test to confirm that subjects are not opioid dependent and a Drug Discrimination Test to ensure that subjects can distinguish between the active control (oxycodone hydrochloride (HCl) immediate-release tablets 40 mg) and placebo.

   Eligible subjects who meet Qualification Criteria will remain as inpatient until the Treatment Phase. Subjects who do not meet Qualification Criteria will be discharged after all post-dose assessments have been performed after the last study drug administration. The last study drug administration in the Qualification Phase and the first study drug administration of the Treatment Phase will be separated by a washout period of approximately 72 hours.
3. Treatment Phase (Visit 2-Continued)

   The Treatment Phase will consist of 5 treatment periods. Subjects will receive each of the following 5 treatments (1 per treatment period) in a randomized, double-blind, crossover manner, following a fasting period of at least 8 hours:
   * Treatment A: PF614 50 mg
   * Treatment B: PF614 100 mg
   * Treatment C: PF614 200 mg
   * Treatment D: Oxycodone IR 40 mg
   * Treatment E: Placebo

   Pharmacodynamic, pharmacokinetic and safety assessments will be conducted prior to dosing and for 24 hours after each study drug administration. Each study drug administration will be separated by a washout interval of approximately 120 hours. All subjects will remain in clinic for the duration of the Treatment Phase. Subjects will be discharged after all post-dose assessments are performed at End of Treatment (EOT), if considered medically suitable for discharge by the investigator.
4. Follow-up Visit (Visit 3) A follow-up visit will be conducted at 8 days (±2 days) after last study drug administration in the Treatment Phase or after early termination (EOS/ET) from the study.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ages 18-55 years, inclusive, in good general health.
* Body mass index (BMI) within the range of 18.0 to 34.0 kg/m2, inclusive, and a minimum weight of 50.0 kg.
* Current opioid users who have used opioids for recreational (non-therapeutic) purposes (i.e., for psychoactive effects) at least 10 times in the past year and have used opioids at least once in the 12 weeks before Screening.
* Must not be physically dependent on opioids, as demonstrated by successful completion of the Naloxone Challenge Test.
* Must meet Drug Discrimination Test (Qualification Phase) eligibility criteria.
* Female subjects must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at admission to Visit 2. Post-menopausal women (i.e., no menstrual period for at least one year) must have a follicle-stimulation hormone (FSH) level >40 milli-international unit (mIU)/mL at Screening.
* Female subjects of child-bearing potential must use an acceptable method of contraception, including abstinence from heterosexual intercourse, hormonal contraceptives, intrauterine device (IUD) with or without hormones, or double-barrier method (e.g., condom and spermicide), for 30 days prior to Screening, during the study and for 30 days following the last administration of study drug.
* Female subjects of non-childbearing potential should be surgically sterile (i.e., have undergone complete hysterectomy, bilateral oophorectomy or tubal ligation) or in a menopausal state (at least 1 year without menses), as confirmed by follicle stimulating hormone (FSH) levels of > 40 IU/L.
* Male subjects must agree to use a double-barrier method (condom and spermicide) or agree to remain abstinent from heterosexual intercourse at the time of screening, during the study and for 90 days following the last administration of study drug.
* Male subjects must agree not to donate sperm during the study and for 90 days following the last administration of study drug.
* Subjects must be able to speak, read, and understand English sufficiently to allow completion of all study assessments.
* Subjects must be able to provide written informed consent.
* Subjects must be willing and able to follow study instructions and be likely to complete all study requirements.

Exclusion Criteria:

* Substance or alcohol dependence (excluding nicotine and caffeine) within the past 2 years, as defined by the Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition - Text Revision (DSM-IV-TR) or a lifetime history of opioid dependence.
* Has ever participated or plans to participate in a substance or alcohol rehabilitation program to treat their substance or alcohol dependence. If participation in a rehabilitation program was court mandated as part of a plea agreement, entry may be permissible at an investigator's discretion.
* Positive urine drug screen (UDS) for substances of abuse at admission to the Qualification Phase, excluding for tetrahydrocannabinol (THC). If a subject presents with a positive UDS at any visit, the subject may be rescheduled or the UDS may be repeated at the discretion of an investigator. If tetrahydrocannabinol (THC) is positive, inclusion will be at the discretion of an investigator, as long as the investigator determines there is no acute intoxication upon presentation.
* History or presence of clinically significant abnormality as assessed by physical examination, medical history, electrocardiograms (ECGs), vital signs, or laboratory values, which, in the opinion of an investigator, would jeopardize the safety of the subject or the validity of the study results. Retesting may be permitted at the discretion of an investigator.
* History or presence of acute respiratory depression, chronic pulmonary disease, cor pulmonale, delirium tremens, central nervous system (CNS) depression or increased cerebrospinal or intracranial pressure.
* Documented history of, or currently active, seizure disorder (excluding febrile seizures in childhood), history of clinically significant head injury or syncope of unknown origin.
* History of gastrointestinal disturbance requiring frequent use of antacids.
* History of or presence of trypsin deficiency.
* Subjects with any history of suicidal ideation within the past 6 months or a lifetime history of suicidal behavior, as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) (baseline version).
* Heavy smoker (>20 cigarettes per day) and/or is unable to abstain from smoking or use of prohibited nicotine-containing products for at least 1 hour before and 8 hours after study drug administration in the Qualification and Treatment Phases (including e-cigarettes, pipes, cigars, chewing tobacco, nicotine topical patches, nicotine gum or nicotine lozenges).
* History of allergy or hypersensitivity to oxycodone, any other opioid or naloxone.
* Female subjects who are currently pregnant (have a positive pregnancy test) or lactating, or who are planning to become pregnant within 30 days of last study drug administration.
* Positive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV).
* Positive result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at check-in to the Qualification Phase (Day -1).
* Evidence of clinically significant hepatic or renal impairment including alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5 × the upper limit of normal (ULN). Retesting may be permitted at the discretion of an investigator.
* Donation or loss of more than 500 mL whole blood within 56 days preceding entry into the Treatment Phase or has donated plasma within 7 days prior to Screening.
* Difficulty with venous access or is unsuitable or unwilling to undergo catheter insertion.
* Use of a prohibited medication or investigational product.
* Is an employee of the sponsor, a research site staff member directly affiliated with this study, or is an immediate family member, defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Any other condition that, in an investigator's opinion, (i) puts the subject at increased risk, (ii) could confound the study results, (iii) may interfere significantly with the subject's participation in the study, or (iv) has the potential to limit the subject's ability to complete the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Peak Maximum Effect (Emax) for Drug Liking (At this Moment) Visual Analog Scale (VAS) | Up to 24 hour post-dose (up to Day 2)
  Relative abuse potential of PF614 compared to Oxycodone and Placebo (I). Emax for drug liking VAS will be reported. Drug liking VAS is a bipolar scale designed to assess a participant's liking for a given study intervention at the time the question is being asked (that is, at this moment). It is scored as an integer ranging from 0 (strong disliking) to 100 (strong liking).
Take Drug Again VAS (Emax) | 12 hours post-dose
  Relative abuse potential of PF614 compared to Oxycodone and Placebo (II). Emax for take drug again VAS will be reported. Peak effect for take drug again based on bipolar VAS from 0 (definitely no) to 100 (definitely so).
Take Drug Again VAS (Emax) | 24 hours post-dose
  Relative abuse potential of PF614 compared to Oxycodone and Placebo (II). Emax for take drug again VAS will be reported. Peak effect for take drug again based on bipolar VAS from 0 (definitely no) to 100 (definitely so).

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Up to 24 hour post-dose (up to Day 2)
  Compare the peak plasma concentration of oxycodone derived from PF614 and oxycodone derived from oxycodone IR tablets
Time to Peak Plasma Concentration (Tmax) | Up to 24 hour post-dose (up to Day 2)
  Compare the time to peak plasma concentration of oxycodone derived from PF614 and oxycodone derived from oxycodone IR tablets
Area Under the Curve Plasma Concentration (AUC 0-24) | Up to 24 hour post-dose (up to Day 2)
  Compare the 0-24 hr pharmacokinetic profile of oxycodone derived from PF614 and oxycodone derived from oxycodone IR tablets
Adverse events (AEs) | Through study completion, an average of 2.5 months
  Safety
Serious adverse events (SAEs) | Through study completion, an average of 2.5 months
  Safety
AEs leading to discontinuation | Through study completion, an average of 2.5 months
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Kirkpatrick, PhD, Study Chair — Ensysce Biosciences
Locations (1):
- Dr. Vince Clinical Research, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan for sharing individual participant data.

REFERENCES:
- [Background] Kirkpatrick DL, Evans C, Pestano LA, Millard J, Johnston M, Mick E, Schmidt WK. Clinical evaluation of PF614, a novel TAAP prodrug of oxycodone, versus OxyContin in a multi-ascending dose study with a bioequivalence arm in healthy volunteers. Clin Transl Sci. 2024 Mar;17(3):e13765. doi: 10.1111/cts.13765. PMID 38511523
- [Background] Kirkpatrick DL, Schmidt WK, Morales R, Cremin J, Seroogy J, Husfeld C, Jenkins T. In vitro and in vivo assessment of the abuse potential of PF614, a novel BIO-MD prodrug of oxycodone. J Opioid Manag. 2017 Jan/Feb;13(1):39-49. doi: 10.5055/jom.2017.0366. PMID 28345745